CLINICAL TRIAL: NCT03796338
Title: Sleep Quantity and Quality in the ICU: a Prospective Observational Study
Brief Title: Sleep Quantity and Quality in the ICU: a Prospective Observational Stud
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, M.D., Careggi Hospital
Other Study IDs: CEAVC, 8611/2018; 11535/OSS
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Sleep Disturbance; Critical Illness
Keywords: intensive care unit; Sleep interruption; Sleep phases
MeSH Terms: conditions — Parasomnias; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Critically ill patients: age > 18 years
  Interventions: Device: Sleep Profiler

INTERVENTIONS:
Device: Sleep Profiler — Patients are observed through a Sleep profiler, routinely used in the intensive care unit (ICU). This device is applied at every patient in the ICU and it acquires EEG, electrooculography, and electromyography from three frontopolar EEG signals.

SUMMARY:
Several evidences in the literature suggest sleep interruption in critical care patients. Nowadays, the amount and the quality of sleep phases during the length of stay in the intensive care unit are largely unknown.

In this study, the amount of time spent by the patients in N1, N2 N3 and REM phases during sleep is quantified.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years

Exclusion Criteria:

* Pregnancy
* Previous enrollment in the same study (sleep recording during previous night)
* Previous use of hypnotic drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Sleep N2 phase | The sleep architecture will be observed during the first night spent in the ICU
  describe the percentage of the total sleep time spent by the patient in N2 stage

SECONDARY OUTCOMES:
Sleep N1 phase | The sleep architecture will be observed during the first night spent in the ICU
  describe the percentage of the total sleep time spent by the patient in N1 stage
Sleep N3 phase | The sleep architecture will be observed during the first night spent in the ICU
  describe the percentage of the total sleep time spent by the patient in N3 stage
Sleep REM phase | The sleep architecture will be observed during the first night spent in the ICU
  describe the percentage of the total sleep time spent by the patient in REM stage

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Villa, MD, Study Director — Azienda Careggi
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No